CLINICAL TRIAL: NCT05715801
Title: The Effects of Hyperbaric Oxygen Therapy on Brain Function in Patients With Cognitive Decline After COVID-19 Infection.
Brief Title: Hyperbaric Oxygen Therapy Improves Brain Function in Patients With Cognitive Decline After COVID-19 Infection.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-KLS-018-01
Record Dates: First submitted 2023-02-01; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Decline; COVID-19; SARS CoV 2 Infection
MeSH Terms: conditions — Cognitive Dysfunction; COVID-19 | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperbaric oxygen therapy (Experimental): Ten sessions of hyperbaric oxygen therapy were completed within 4 weeks of enrollment.
  Interventions: Procedure: hyperbaric oxygen therapy
- conventional oxygen therapy (Active Comparator): Ten sessions of conventional oxygen therapy were completed within 4 weeks after enrollment.
  Interventions: Procedure: conventional oxygen therapy

INTERVENTIONS:
Procedure: hyperbaric oxygen therapy — The hyperbaric oxygen group was given 60 minutes of pure oxygen under 2ATA (Atmosphere Absolute, ATA) and 5 minutes of rest in between.
  Arms: hyperbaric oxygen therapy
Procedure: conventional oxygen therapy — Conventional oxygen therapy group breathed 27% oxygen at 1.03 ATA for 60 minutes. (The chamber pressure was increased to 1.2ATA with circulating air noise for the first 5 minutes of the experiment, then reduced to 1.03 ATA for the next 5 minutes.)
  Arms: conventional oxygen therapy

SUMMARY:
COVID-19 has swept the world, and while some people may experience long-term cognitive decline as a result of infection, no effective treatment has been announced. The primary goal of this study was to determine the efficacy of hyperbaric oxygen therapy in patients with SARS-CoV-2 infection, as well as to assess the effect of hyperbaric oxygen therapy on brain function in patients with COVID-19-related cognitive decline. In this study, approximately 80 people were randomly assigned to either hyperbaric oxygen or regular oxygen therapy to compare the effects of these two treatments on disease.

DETAILED DESCRIPTION:
80 patients with cognitive impairment following a novel coronavirus infection will be randomly assigned to one of two treatment groups: hyperbaric oxygen therapy or conventional oxygen therapy.

After the intervention, the improvement of hyperbaric oxygen on cognition, fatigue, sleep disorders, anxiety and depression, and other clinical manifestations was observed. The neurologic function of hyperbaric oxygen in the treatment of patients with cognitive decline after SARS-CoV-2 infection was also evaluated from imaging and electrophysiological multi-dimensional indexes.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients 4 weeks after the diagnosis of SARS-CoV-2 infection
* Subjective cognitive decline after SARS-CoV-2 infection
* SARS-CoV-2 nucleic acid/antigen test negative.

Exclusion Criteria:

* Contraindications to hyperbaric oxygen therapy
* Cognitive decline can be explained by other diseases
* Conditions that researchers consider unsuitable for clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-29 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
scores of Montreal Cognitive Scale (MoCA) | The patients would be followed up for 3 months after oxygen therapy.
  The total score is 30 points, and the cut-off value for MCI is identified:≤19 points(illiterate and primary school group);≤22 points(Middle school group); ≤24 points(University group).

SECONDARY OUTCOMES:
Quantitative Electroencephalography | The patients would be followed up for 3 months after oxygen therapy.
  The main frequency distribution and absolute power spectrum of 4 frequency bands (δ (1-3.9 Hz) , θ (4-7 Hz) , α (8-12.9 Hz) and β (13-30 Hz) were obtained, the θ frequency and the relative power of δ frequency (DTABR = (δ + θ)/(α + β)) were calculated.
Brain magnetic resonance imaging (MRI), brain functional magnetic resonance imaging (fMRI) | The patients would be followed up for 3 months after oxygen therapy.
  The time series acquired from resting-state fMRI will be transformed into the frequency domain using Fast Fourier transform, and the square root of the power spectrum will be calculated and averaged across 0.01-0.08 Hz within each voxel.The ALFF of each voxel will be divided by the global mean ALFF value to standardize data across subjects.
Boston naming test | The patients would be followed up for 3 months after oxygen therapy.
  Total score is 30 points.The cut-off values for each group are:≦19(Junior high school education level),≦21(High school education level),≦22(University education level)
auditory verbal learning test，AVLT | The patients would be followed up for 3 months after oxygen therapy.
  A 12-word list was repeated 3 times, and short-delayed recall was performed after an interval of 3-5 minutes, and long-delayed recall, cued recall and recognition were performed after an interval of 20 minutes. The most sensitive evaluation indexes were long-delayed recall score and recognition score. The auxiliary indexes included immediate recall score, total recall score, recall skills and discrimination. Cut-off values: long delayed recall score ≤5 (50-59 years), ≤4 (60-69 years), ≤3 (70-79 years);Recognition score ≤20 (50-59 years), ≤19 (60-69 years), ≤18 (70-79 years).
The Shape Trail Making Test A and B(STT-A&B) | The patients would be followed up for 3 months after oxygen therapy.
  The Shape Trail Making Test A and B(STT-A&B) is divided into two parts: A and B. Each part includes exercises and tests. Part A asks participants to connect random numbers in sequence as quickly as possible. Part B asks participants to connect numbers in sequence alternately. Rating: Mainly record the amount of time spent. Cut-off value: STT-A test questions, 50~59 years old ≥70s, 60~69 years old ≥80s, 70~79 years old ≥100s;STT-B test questions, 50~59 years old ≥180s, 60~69 years old ≥200s, 70~79 years old ≥240s. The longer it takes, the worse it gets.
Animal word fluency (AFT) | The patients would be followed up for 3 months after oxygen therapy.
  Subjects were asked to list as many examples of animals as possible within 1 min. Cut-off value: animal fluency score ≤12(junior high school group) , ≤13(senior high school group) , ≤14(university group)
Stroop color words test | The patients would be followed up for 3 months after oxygen therapy.
  The stroop test lasts for 45 seconds, and the correct number of each test is calculated.Cut-off value: animal fluency score ≤12(junior high school group) , ≤13(senior high school group) , ≤14(university group)

CONTACTS AND LOCATIONS:
Overall Officials: Jiannong Wu, M.D., Study Chair — First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided